CLINICAL TRIAL: NCT05197400
Title: A Prospective Randomized Comparison of the Effect of Supine and Prone Position on the Ultrasonographic Upper Airway Measurements and Postoperative Critical Respiratory Events
Brief Title: Comparison of the Effect of Supine and Prone Position on the Ultrasonographic Airway Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Işıl Karabeyoğlu, anaestesia and reanimation, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: E1-21-2261
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2023-01

CONDITIONS: Airway Edema; Obstructive Sleep Apnea; Respiratory Complication
Keywords: airway edema; obstructive sleep apnea; respiratory complications
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- supine (Active Comparator): operation in the supine position
  Interventions: Diagnostic Test: preoperative airway ultrasonography; Diagnostic Test: postoperative airway ultrasonography
- prone (Active Comparator): operation in the prone position
  Interventions: Diagnostic Test: preoperative airway ultrasonography; Diagnostic Test: postoperative airway ultrasonography

INTERVENTIONS:
Diagnostic Test: preoperative airway ultrasonography — Tongue thickness Median sagittal tongue cross-sectional area Tongue width
  Tongue volume:
  Lateral parapharyngeal wall thickness
Diagnostic Test: postoperative airway ultrasonography — Tongue thickness Median sagittal tongue cross-sectional area Tongue width
  Tongue volume:
  Lateral parapharyngeal wall thickness

SUMMARY:
The aim of this study is to compare the preoperative and postoperative ultrasonographic measurements of patients undergoing in the prone position and the change in upper airway edema.

The secondary aim of the study is to investigate the relationship between OSAS risk levels determined by the STOP-BANG score in the preoperative period of the patients participating in the study, and airway ultrasound measurements and postoperative critical respiratory events in the preoperative and postoperative period.

ELIGIBILITY:
Inclusion Criteria:1-American Society of Anesthesiologists Physical Status Classification (ASA) I-II-III-IV risk group who will undergo Percutaneous Nephrolithotomy surgery

Exclusion Criteria:

1. prone position contraindications
2. history of maxillofacial deformity, tumor or trauma,
3. difficult airway history
4. decompensated cardiac, respiratory, hepatic, renal diseases
5. cervical spine fracture
6. Patients refusal -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Preoperative Tongue thickness | Baseline, preoperative
postoperative Tongue thickness1 | postextubation
postoperative Tongue thickness2 | postoperative 2. hour]
preoperative Tongue volume | Baseline, preoperative
postoperative Tongue volume1 | postextubation
postoperative Tongue volume2 | postoperative 2. hour
Preoperative Lateral parapharyngeal wall thickness | Baseline, preoperative
postoperative Lateral parapharyngeal wall thickness1 | postextubation
postoperative Lateral parapharyngeal wall thickness2 | postoperative 2. hour
Critical respiratory events | Within postoperative 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: ışıl karabeyoğlu, md, Principal Investigator — ankara ch bilkent; betül güven aytaç, Study Chair — Ankara CH bilkent
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No